CLINICAL TRIAL: NCT03485898
Title: Patient Outcomes After an Hospitalization in the Specialized Cognitive-behavioral Unit (UCC) of Toulon
Brief Title: Study of Patients Hospitalized in Specialized Cognitive-behavioral Unit (UCC)
Acronym: UCC
Status: Terminated | Type: Observational
Why Stopped: study director job transfer in another departement
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-CHITS-05; 2017-A03332-51 (Other: Id-RCB)
Record Dates: First submitted 2018-02-22; First posted 2018-04-03 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Behavior Disorders
Keywords: UCC; mortality; alzheimer's disease; longitudinal study
MeSH Terms: conditions — Mental Disorders; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to assess the mortality of patient discharged from the specialized cognitive-behavioral unit (UCC) of Toulon.

DETAILED DESCRIPTION:
The purpose of specialized cognitive-behavioral unit is to take care of patients demented, valid and with disruptive behavior disorders. The hypothesis is that analyzing the healthcare of these discharged patients might provide a view of the benefices of these units.

The study will be explained to the eligible subjects if they are able to understand it, or to their trusted person, primary caregiver or legal representative.

Medical information will be collected during and after the hospitalization in the specialized cognitive-behavioral unit. The investigator will call the medical staff and the primary caregiver at 3, 6, and 12 months after the patient's discharge, in order to collect study data.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at the UCC of Toulon

Exclusion Criteria:

* Patient already included in the study ( a patient cannot be included twice during the study)
* Non-affiliated to a social security regimen
* Objection of the patient, the trusted person, the legal representative, the relative or the member of the family (depending on the overall condition of the patient)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population correspond to all inpatient from the UCC of Toulon
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Mortality rate at 12 month after patient's discharge from UCC | 12 months
  Number of dead patient at 12 month on the total number of patient included

SECONDARY OUTCOMES:
Mortality rate at 3 and 6 month after patient's discharge from UCC | 3 and 6 months
  Number of dead patient at 3 and 6 month on the total number of patient included
Assess the primary mortality risk factors regarding all the collected data. | 12 months
  correlation analysis of collected data and survival data will lead to prediction of survival model with the most relevant survival variable
Create a predictive score for 6 and 12 month mortality | 6 and 12 months
  all the survival variable will have a score according to the survival prediction model - this endpoint is adressed in order to create a predictive scale/score.
Mortality rate during the hospitalization in the UCC | 12 months
  Number of all dead patient on the total number of patient included
Analysis of hospitalisation rate | 12 months
  Descriptive analysis
Analysis of the number of treatment taken during the study | 12 months
  Descriptive analysis
Analysis of the different classes of treatment taken during the study | 12 months
  Descriptive analysis of the rate of different classes of treatment taken by patient during the study
Analysis of the treatment's mode of delivery | 12 months
  Descriptive analysis

CONTACTS AND LOCATIONS:
Overall Officials: Romain Van overloop, doctor, Principal Investigator — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal de Toulon La-Seyne-sur-Mer, Toulon, France

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Walsh JS, Welch HG, Larson EB. Survival of outpatients with Alzheimer-type dementia. Ann Intern Med. 1990 Sep 15;113(6):429-34. doi: 10.7326/0003-4819-113-6-429. PMID 2386336
- [Background] Molsa PK, Marttila RJ, Rinne UK. Survival and cause of death in Alzheimer's disease and multi-infarct dementia. Acta Neurol Scand. 1986 Aug;74(2):103-7. doi: 10.1111/j.1600-0404.1986.tb04634.x. PMID 3776457
- [Background] Edland SD, Rocca WA, Petersen RC, Cha RH, Kokmen E. Dementia and Alzheimer disease incidence rates do not vary by sex in Rochester, Minn. Arch Neurol. 2002 Oct;59(10):1589-93. doi: 10.1001/archneur.59.10.1589. PMID 12374497
- [Background] Fitzpatrick AL, Kuller LH, Lopez OL, Kawas CH, Jagust W. Survival following dementia onset: Alzheimer's disease and vascular dementia. J Neurol Sci. 2005 Mar 15;229-230:43-9. doi: 10.1016/j.jns.2004.11.022. Epub 2004 Dec 23. PMID 15760618
- [Background] Lee M, Chodosh J. Dementia and life expectancy: what do we know? J Am Med Dir Assoc. 2009 Sep;10(7):466-71. doi: 10.1016/j.jamda.2009.03.014. Epub 2009 Jun 27. PMID 19716062
- [Background] Mitchell SL, Kiely DK, Hamel MB, Park PS, Morris JN, Fries BE. Estimating prognosis for nursing home residents with advanced dementia. JAMA. 2004 Jun 9;291(22):2734-40. doi: 10.1001/jama.291.22.2734. PMID 15187055
- [Background] Mitchell SL, Miller SC, Teno JM, Davis RB, Shaffer ML. The advanced dementia prognostic tool: a risk score to estimate survival in nursing home residents with advanced dementia. J Pain Symptom Manage. 2010 Nov;40(5):639-51. doi: 10.1016/j.jpainsymman.2010.02.014. PMID 20621437
- [Background] Mitchell SL, Miller SC, Teno JM, Kiely DK, Davis RB, Shaffer ML. Prediction of 6-month survival of nursing home residents with advanced dementia using ADEPT vs hospice eligibility guidelines. JAMA. 2010 Nov 3;304(17):1929-35. doi: 10.1001/jama.2010.1572. PMID 21045099